CLINICAL TRIAL: NCT03694197
Title: Long Term Safety Study of PRALUENT in Patients With Heterozygous Familial Hypercholesterolemia or With Non-Familial Hypercholesterolemia at High and Very High Cardiovascular Risk and Previously Enrolled in the Neurocognitive Function Trial
Brief Title: Long Term Safety Study of PRALUENT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The primary objective (to evaluate the long-term safety of Praluent) was adequately evaluated in other studies.
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R727-CL-1609; 2018-002810-11 (EudraCT Number)
Record Dates: First submitted 2018-09-06; First posted 2018-10-03 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Heterozygous Familial Hypercholesterolemia; Non-familial Hypercholesterolemia
MeSH Terms: interventions — alirocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label (Experimental)
  Interventions: Drug: Praluent

INTERVENTIONS:
Drug: Praluent — Subcutaneous (SC) administration
  Other Names: Alirocumab; REGN727; SAR236553

SUMMARY:
The primary objective of the study was to evaluate the long term safety of PRALUENT in participants with heterozygous familial hypercholesterolemia (heFH) or non-familial hypercholesterolemia (FH) participants at high or very high cardiovascular risk who completed the neurocognitive function study R727-CL-1532 (NCT02957682).

The secondary objectives of the study were:

* To evaluate the effect of PRALUENT on low-density lipoprotein cholesterol (LDL-C)
* To evaluate the effect of PRALUENT on other lipid parameters
* To evaluate the effect of PRALUENT on gonadal steroid hormones

ELIGIBILITY:
Key Inclusion Criteria:

Participants randomized into the neurocognitive function study (R727-CL-1532) who completed treatment and the end of study (EOS) visit with no premature or permanent discontinuation of study drug.

Key Exclusion Criteria:

1. Significant protocol deviation in the parent study (neurocognitive function study R727-CL-1532: NCT02957682) based on the investigator's or sponsor's judgment, such as noncompliance
2. Any participant who experienced an AE leading to permanent discontinuation from the neurocognitive function study R727-CL-1532 (NCT02957682).
3. Any new condition or worsening of an existing condition which, in the opinion of the investigator or per the PRALUENT local label, would make the participant unsuitable for enrollment or could interfere with the participant participating in or completing the open-label extension (OLE) study
4. Known hypersensitivity to monoclonal antibody or any component of the drug product
5. Pregnant or breastfeeding women

Note: Other inclusion/ exclusion criteria apply

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1389 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (105):
- United States (55):
  - Regeneron Research Site, Auburn, Alabama
  - Regeneron Research Site, Mobile, Alabama
  - Regeneron Research Site, Beverly Hills, California
  - Regeneron Research Site, Los Gatos, California
  - Regeneron Research Site, North Hollywood, California
  - Regeneron Research Site, Port Hueneme, California
  - Regeneron Research Site, Aurora, Colorado
  - Regeneron Research Site, Colorado Springs, Colorado
  - Regeneron Research Site, Lake Worth, Florida
  - Regeneron Research Site, Miami Springs, Florida
  - Regeneron Research Site, Champaign, Illinois
  - Regeneron Research Site, Evansville, Indiana
  - Regeneron Research Site, Indianapolis, Indiana
  - Regeneron Research Site, Ames, Iowa
  - Regeneron Research Site, Iowa City, Iowa
  - Regeneron Research Site, Waterloo, Iowa
  - Regeneron Research Site, Newton, Kansas
  - Regeneron Research Site, Louisville, Kentucky
  - Regeneron Research Site, Bangor, Maine
  - Regeneron Research Site, Baltimore, Maryland
  - Regeneron Research Site, Oxon Hill, Maryland
  - Regeneron Research Site, Olive Branch, Mississippi
  - Regeneron Research Site, Washington, Missouri
  - Regeneron Research Site, Buffalo, New York
  - Regeneron Research Site, New Hyde Park, New York
  - Regeneron Research Site, Cary, North Carolina
  - Regeneron Research Site, Charlotte, North Carolina
  - Regeneron Research Site, Greensboro, North Carolina
  - Regeneron Research Site, Hickory, North Carolina
  - Regeneron Research Site, Raleigh, North Carolina
  - Regeneron Research Site, Rocky Mount, North Carolina
  - Regeneron Research Site, Salisbury, North Carolina
  - Regeneron Research Site, Statesville, North Carolina
  - Regeneron Research Site, Wilmington, North Carolina
  - Regeneron Research Site, Winston-Salem, North Carolina
  - Regeneron Research Site, Cincinnati, Ohio
  - Regeneron Research Site, Cleveland, Ohio
  - Regeneron Research Site, Dayton, Ohio
  - Regeneron Research Site, Charleston, South Carolina
  - Regeneron Research Site, Summerville, South Carolina
  - Regeneron Research Site, Rapid City, South Dakota
  - Regeneron Research Site, Bristol, Tennessee
  - Regeneron Research Site 2, Knoxville, Tennessee
  - Regeneron Research Site 3, Knoxville, Tennessee
  - Regeneron Research Site, Knoxville, Tennessee
  - Regeneron Research Site, Powell, Tennessee
  - Regeneron Research Site, Dallas, Texas
  - Regeneron Research Site, Houston, Texas
  - Regeneron Research Site, Schertz, Texas
  - Regeneron Research Site, Shavano Park, Texas
  - Regeneron Research Site, Falls Church, Virginia
  - Regeneron Research Site, Winchester, Virginia
  - Regeneron Research Site, Tacoma, Washington
  - Regeneron Research Site, Walla Walla, Washington
  - Regeneron Research Site, Manitowoc, Wisconsin
- Bulgaria (6):
  - Regeneron Research Site, Pleven
  - Regeneron Research Site, Plovdiv
  - Regeneron Research Site, Sofia
  - Regeneron Research Site #2, Sofia
  - Regeneron Research Site, Stara Zagora
  - Regeneron Research Site, Varna
- Estonia (5):
  - Regeneron Research Site, Tallinn, Harju
  - Regeneron Research Site, Paide
  - Regeneron Research Site #2, Tallinn
  - Regeneron Research Site, Tallinn
  - Regeneron Research Site, Tartu
- Russia (13):
  - Regeneron Research Site, Ivanovo
  - Regeneron Research Site, Kirov
  - Regeneron Research Site, Moscow
  - Regeneron Research Site, Novosibirsk
  - Regeneron Research Site, Rostov-on-Don
  - Regeneron Research Site #2, Saint Petersburg
  - Regeneron Research Site, Saint Petersburg
  - Regeneron Research Site, Saratov
  - Regeneron Research Site, Sverdlovskaya
  - Regeneron Research Site, Tyumen
  - Regeneron Research Site 1, Yaroslavl
  - Regeneron Research Site 2, Yaroslavl
  - Regeneron Research Site, Yekaterinburg
- South Africa (16):
  - Regeneron Research Site, Kuilsrivier, Cape Town
  - Regeneron Research Site, Parow, Cape Town
  - Regeneron Research Site, Port Elizabeth, Eastern Cape
  - Regeneron Research Site, Halfway House, Gauteng
  - Regeneron Research Site, Pretoria, Gauteng
  - Regeneron Research Site, Pretoria West, Gauteng
  - Regeneron Research Site, Kempton Park, Johannesburg
  - Regeneron Research Site, Soweto, Johannesburg
  - Regeneron Research Site, Cape Town, Western Cape
  - Regeneron Research Site, George, Western Cape
  - Regeneron Research Site, Paarl, Western Cape
  - Regeneron Research Site, Somerset West, Western Cape
  - Regeneron Research Site, Worcester, Western Cape
  - Regeneron Research Site, Bloemfontein
  - Regeneron Research Site, Claremont
  - Regeneron Research Site, Johannesburg
- Ukraine (10):
  - Regeneron Research Site #2, Kharkiv
  - Regeneron Research Site, Kharkiv
  - Regeneron Research Site, Kiev
  - Regeneron Research Site, Kyiv
  - Regeneron Research Site #2, Kyiv
  - Regeneron Research Site, Lviv
  - Regeneron Research Site, Uzhhorod
  - Regeneron Research Site, Vinnitsa
  - Regeneron Research Site, Vinnitsya
  - Regeneron Research Site, Vinnytsia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The 1389 participants who completed double-blind treatment and the end-of-study (EOS) visit in R727-CL-1532 (NCT02957682) signed consent and were screened for this open-label study (EOS visit corresponded to day 1/visit 1 of this study).
Pre-assignment Details: First subcutaneous (SC) injection was administered in the clinic (day 1/visit 1). Four of the1389 participants discontinued on day 1 before treatment: 2 discontinued due to failure to meet inclusion/exclusion criteria,1 withdrew consent, and 1 discontinued due to adverse event (AE). A total of 1385 participants received any study drug on day 1.
Groups:
- Alirocumab 75 Q2W/Up150 Q2W: All participants initiated treatment with PRALUENT (alirocumab) at the starting dose of 75 milligrams (mg) once every 2 weeks (Q2W). After week 8, the dose could be adjusted (up to 150 mg Q2W, maintained or from 150 mg Q2W to 75 mg Q2W) if needed based on low-density lipoprotein cholesterol (LDL-C) levels.
Period: Overall Study
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Started (Safety analysis set (SAF): all participants who received any study drug) | 1385
Completed (The study was terminated early by the Sponsor before any participants completed the originally planned treatment period of up to 192 weeks.) | 0
Not Completed | 1385
Not completed — Adverse Event | 9
Not completed — Protocol became inconvenient to participate | 1
Not completed — Physician Decision | 4
Not completed — Study terminated by sponsor | 1350
Not completed — Participant moved | 5
Not completed — Participant withdrew consent | 10
Not completed — Related to IMP administration | 1
Not completed — Not disclosed | 5

BASELINE CHARACTERISTICS:
Population: Demographic and other baseline characteristics were based on the data collected in R727-CL-1532 (NCT02957682). The baseline value was generally defined as the last available value before the first dose of double-blind study treatment in that study.
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 527
  Male | 858
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 1372
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 1178
    Black or African American | 81
    Asian | 7
    American Indian or Alaska Native | 1
    Native Hawaiian or Other Pacific Islander | 0
    Other | 118

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE) After First Administration of Study Drug Through the Last Dose of Study Drug Plus 2 Weeks
Description: An AE is any untoward medical occurrence in a participant administered a study drug which may or may not have a causal relationship with the study drug. AEs include serious adverse events (SAEs), AEs leading to treatment discontinuation, and adverse events of special interest (AESI). AESI include local injection site reactions, general allergic events, elevated alanine aminotransferase (ALT) levels greater than or equal to (≥) 3 upper limit normal (ULN) (if baseline is less than (<) ULN)/ALT ≥2 x ULN (if baseline ≥ ULN), neurologic events, neurocognitive events (according to Customized Medical Dictionary for Regulatory Activities [MedDRA] Query [CMQ] by Sponsor grouping and CMQ by FDA grouping), cataract, new onset diabetes (NOD), hepatic disorders, and diabetes mellitus (DM)/diabetic complications.
Time Frame: After first administration of study drug through the last dose of study drug plus 2 weeks, up to 80 weeks
Population: Safety analysis set (SAF): All participants who received any study drug
Measure: Number; unit: Participants
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
Participants
  Any treatment emergent adverse event (TEAE) | 568
  Any treatment emergent serious adverse event (SAE) | 89
  Any TEAE leading to death | 5
  Any TEAE leading to permanent treatment discontinuation | 9
  Any neurocognitive disorders TEAE (by Sponsor CMQ) | 4
  Any neurocognitive disorders TEAE (by FDA CMQ) | 0
  Any NOD; # analyzed = # of participants w/out diabetes at baseline: number analyzed (Participants) | 687
  Any NOD; # analyzed = # of participants w/out diabetes at baseline | 15
  Any hepatic disorders TEAE | 14
  Any neurological TEAE | 15
  Any general allergic TEAE | 25
  At least one treatment-emergent injection site reaction | 22
  Any cataract TEAE | 5
  Any elevated ALT ≥3 ULN: number analyzed (Participants) | 1305
  Any elevated ALT ≥3 ULN | 1
  Any DM/diabetic complications TEAE; # analyzed = # of participants w/diabetes at baseline: number analyzed (Participants) | 698
  Any DM/diabetic complications TEAE; # analyzed = # of participants w/diabetes at baseline | 41
  Any DM/diabetic complications TEAE; # analyzed = # of participants w/out diabetes at baseline: number analyzed (Participants) | 687
  Any DM/diabetic complications TEAE; # analyzed = # of participants w/out diabetes at baseline | 3

2. Secondary Outcome: Calculated Low-density Lipoprotein Cholesterol (LDL-C) Values From Baseline Over Time
Description: The baseline value was defined as the last available value before the first dose of double-blind study treatment in study R727-CL-1532 (NCT02957682)
Time Frame: Up to week 72
Population: SAF (All participants who received any study drug); Here, "Number Analyzed" = Number of participants evaluable at that timepoint
Measure: Mean (Standard Deviation); unit: Milligrams per decilitre (mg/dL)
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
Milligrams per decilitre (mg/dL)
  Baseline: number analyzed (Participants) | 1367
  Baseline | 117.8 (40.67)
  Week 8: number analyzed (Participants) | 1345
  Week 8 | 58.9 (37.31)
  Week 12: number analyzed (Participants) | 356
  Week 12 | 63.6 (40.79)
  Week 24: number analyzed (Participants) | 769
  Week 24 | 56.2 (36.59)
  Week 48: number analyzed (Participants) | 311
  Week 48 | 56.8 (36.13)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 52.2 (38.80)

3. Secondary Outcome: Percent Change in LDL-C From Baseline Over Time
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
Percent Change
  Week 8: number analyzed (Participants) | 1328
  Week 8 | -48.74 (31.121)
  Week 12: number analyzed (Participants) | 353
  Week 12 | -44.64 (35.338)
  Week 24: number analyzed (Participants) | 754
  Week 24 | -50.75 (30.249)
  Week 48: number analyzed (Participants) | 301
  Week 48 | -52.35 (27.929)
  Week 72: number analyzed (Participants) | 54
  Week 72 | -51.21 (32.742)

4. Secondary Outcome: Total Cholesterol (Total-C) Values From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
mg/dL
  Baseline | 199.5 (48.88)
  Week 8: number analyzed (Participants) | 1346
  Week 8 | 139.5 (44.76)
  Week 12: number analyzed (Participants) | 356
  Week 12 | 145.0 (48.68)
  Week 24: number analyzed (Participants) | 769
  Week 24 | 137.3 (44.18)
  Week 48: number analyzed (Participants) | 311
  Week 48 | 139.5 (44.53)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 131.7 (43.25)

5. Secondary Outcome: Percent Change From Baseline in Total-C Over Time
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
Percent Change
  Week 8: number analyzed (Participants) | 1346
  Week 8 | -28.68 (20.158)
  Week 12: number analyzed (Participants) | 356
  Week 12 | -25.99 (23.058)
  Week 24: number analyzed (Participants) | 769
  Week 24 | -29.98 (20.930)
  Week 48: number analyzed (Participants) | 311
  Week 48 | -30.89 (21.004)
  Week 72: number analyzed (Participants) | 54
  Week 72 | -31.55 (22.238)

6. Secondary Outcome: Lipoprotein a (Lp(a)) Values From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
mg/dL
  Baseline | 39.7 (47.86)
  Week 8: number analyzed (Participants) | 190
  Week 8 | 35.0 (41.99)
  Week 12: number analyzed (Participants) | 353
  Week 12 | 32.7 (39.42)
  Week 24: number analyzed (Participants) | 419
  Week 24 | 33.9 (42.54)
  Week 48: number analyzed (Participants) | 311
  Week 48 | 38.6 (50.66)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 40.4 (56.47)

7. Secondary Outcome: Percent Change From Baseline in Lp(a) Over Time
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
Percent Change
  Week 8: number analyzed (Participants) | 190
  Week 8 | -12.69 (35.452)
  Week 12: number analyzed (Participants) | 353
  Week 12 | 10.63 (228.659)
  Week 24: number analyzed (Participants) | 419
  Week 24 | -6.80 (110.827)
  Week 48: number analyzed (Participants) | 311
  Week 48 | -7.89 (116.831)
  Week 72: number analyzed (Participants) | 54
  Week 72 | -22.23 (28.233)

8. Secondary Outcome: Non-high-density Lipoprotein Cholesterol (Non-HDL-C) Values From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
mg/dL
  Baseline | 152.4 (48.81)
  Week 8: number analyzed (Participants) | 1346
  Week 8 | 88.5 (43.54)
  Week 12: number analyzed (Participants) | 356
  Week 12 | 94.3 (48.77)
  Week 24: number analyzed (Participants) | 769
  Week 24 | 87.3 (43.56)
  Week 48: number analyzed (Participants) | 311
  Week 48 | 88.9 (44.25)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 80.9 (42.67)

9. Secondary Outcome: Percent Change From Baseline in Non-HDL-C Over Time
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
Percent Change
  Week 8: number analyzed (Participants) | 1346
  Week 8 | -40.35 (27.470)
  Week 12: number analyzed (Participants) | 356
  Week 12 | -36.89 (29.567)
  Week 24: number analyzed (Participants) | 769
  Week 24 | -41.47 (26.763)
  Week 48: number analyzed (Participants) | 311
  Week 48 | -42.33 (28.728)
  Week 72: number analyzed (Participants) | 54
  Week 72 | -43.28 (29.534)

10. Secondary Outcome: High-density Lipoprotein Cholesterol (HDL-C) Values From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
mg/dL
  Baseline | 47.1 (13.92)
  Week 8: number analyzed (Participants) | 1346
  Week 8 | 51.0 (14.82)
  Week 12: number analyzed (Participants) | 356
  Week 12 | 50.6 (13.95)
  Week 24: number analyzed (Participants) | 769
  Week 24 | 49.9 (14.80)
  Week 48: number analyzed (Participants) | 311
  Week 48 | 50.5 (14.66)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 50.8 (14.61)

11. Secondary Outcome: Percent Change From Baseline in HDL-C Over Time
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
Percent Change
  Week 8: number analyzed (Participants) | 1346
  Week 8 | 10.54 (22.735)
  Week 12: number analyzed (Participants) | 356
  Week 12 | 10.33 (21.933)
  Week 24: number analyzed (Participants) | 769
  Week 24 | 8.53 (21.824)
  Week 48: number analyzed (Participants) | 311
  Week 48 | 9.81 (23.690)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 9.24 (21.505)

12. Secondary Outcome: Fasting Triglycerides (TGs) Values From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
mg/dL
  Baseline | 179.2 (146.51)
  Week 8: number analyzed (Participants) | 1346
  Week 8 | 154.8 (113.05)
  Week 12: number analyzed (Participants) | 356
  Week 12 | 162.2 (182.00)
  Week 24: number analyzed (Participants) | 769
  Week 24 | 169.3 (161.45)
  Week 48: number analyzed (Participants) | 311
  Week 48 | 171.1 (131.35)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 156.9 (65.21)

13. Secondary Outcome: Percent Change From Baseline in Fasting TGs Over Time
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
Percent Change
  Week 8: number analyzed (Participants) | 1346
  Week 8 | -4.68 (49.230)
  Week 12: number analyzed (Participants) | 356
  Week 12 | -4.29 (40.748)
  Week 24: number analyzed (Participants) | 769
  Week 24 | 0.42 (54.118)
  Week 48: number analyzed (Participants) | 311
  Week 48 | 1.54 (69.156)
  Week 72: number analyzed (Participants) | 54
  Week 72 | -5.97 (41.440)

14. Secondary Outcome: Apolipoprotein B (Apo B) Values From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
mg/dL
  Baseline | 103.8 (27.25)
  Week 8: number analyzed (Participants) | 190
  Week 8 | 62.5 (27.63)
  Week 12: number analyzed (Participants) | 353
  Week 12 | 68.0 (31.32)
  Week 24: number analyzed (Participants) | 420
  Week 24 | 61.5 (26.20)
  Week 48: number analyzed (Participants) | 311
  Week 48 | 63.7 (26.40)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 58.5 (25.82)

15. Secondary Outcome: Percent Change From Baseline in Apo B Over Time
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
Percent Change
  Week 8: number analyzed (Participants) | 190
  Week 8 | -36.51 (34.460)
  Week 12: number analyzed (Participants) | 353
  Week 12 | -34.48 (27.905)
  Week 24: number analyzed (Participants) | 420
  Week 24 | -38.16 (24.867)
  Week 48: number analyzed (Participants) | 311
  Week 48 | -37.93 (23.767)
  Week 72: number analyzed (Participants) | 54
  Week 72 | -39.04 (26.383)

16. Secondary Outcome: Apolipoprotein-A1 (Apo A1) Values From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
mg/dL
  Baseline | 145.3 (24.95)
  Week 8: number analyzed (Participants) | 190
  Week 8 | 148.5 (24.73)
  Week 12: number analyzed (Participants) | 353
  Week 12 | 149.4 (25.38)
  Week 24: number analyzed (Participants) | 420
  Week 24 | 150.7 (26.36)
  Week 48: number analyzed (Participants) | 311
  Week 48 | 152.6 (25.96)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 151.4 (26.03)

17. Secondary Outcome: Percent Change From Baseline in Apo A1 Over Time
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
Percent Change
  Week 8: number analyzed (Participants) | 190
  Week 8 | 5.07 (13.385)
  Week 12: number analyzed (Participants) | 353
  Week 12 | 2.99 (13.638)
  Week 24: number analyzed (Participants) | 420
  Week 24 | 5.35 (14.108)
  Week 48: number analyzed (Participants) | 311
  Week 48 | 4.77 (13.836)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 1.21 (13.170)

18. Secondary Outcome: Gonadal Hormone (Follicle Stimulating Hormone [FSH] and Luteinizing Hormone [LH]) Values for Female Participants From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: SAF (Female participants who received any study drug); Here, "Number Analyzed" = Number of female participants evaluable at that timepoint
Measure: Mean (Standard Deviation); unit: International units per litre (IU/L)
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 527
International units per litre (IU/L)
  FSH Baseline | 57.948 (26.7383)
  FSH Week 8: number analyzed (Participants) | 84
  FSH Week 8 | 59.264 (24.7912)
  FSH Week 12: number analyzed (Participants) | 135
  FSH Week 12 | 54.279 (23.9923)
  FSH Week 24: number analyzed (Participants) | 280
  FSH Week 24 | 57.664 (25.9830)
  FSH Week 48: number analyzed (Participants) | 106
  FSH Week 48 | 56.529 (25.1408)
  FSH Week 72: number analyzed (Participants) | 23
  FSH Week 72 | 58.600 (24.5205)
  LH Baseline | 30.155 (13.1090)
  LH Week 8: number analyzed (Participants) | 84
  LH Week 8 | 33.794 (14.4459)
  LH Week 12: number analyzed (Participants) | 135
  LH Week 12 | 30.779 (13.0946)
  LH Week 24: number analyzed (Participants) | 280
  LH Week 24 | 31.260 (13.7344)
  LH Week 48: number analyzed (Participants) | 106
  LH Week 48 | 29.585 (13.9792)
  LH Week 72: number analyzed (Participants) | 23
  LH Week 72 | 29.248 (11.0829)

19. Secondary Outcome: Change From Baseline in Gonadal Hormones (FSH and LH) for Female Participants Over Time
Time Frame: Up to week 72
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 527
IU/L
  FSH Week 8: number analyzed (Participants) | 84
  FSH Week 8 | -0.765 (12.0083)
  FSH Week 12: number analyzed (Participants) | 135
  FSH Week 12 | -0.984 (12.1584)
  FSH Week 24: number analyzed (Participants) | 280
  FSH Week 24 | -0.575 (8.7780)
  FSH Week 48: number analyzed (Participants) | 106
  FSH Week 48 | -0.877 (15.9972)
  FSH Week 72: number analyzed (Participants) | 23
  FSH Week 72 | -1.861 (8.6119)
  LH Week 8: number analyzed (Participants) | 84
  LH Week 8 | 2.730 (8.2258)
  LH Week 12: number analyzed (Participants) | 135
  LH Week 12 | 1.882 (8.2884)
  LH Week 24: number analyzed (Participants) | 280
  LH Week 24 | 0.939 (6.3694)
  LH Week 48: number analyzed (Participants) | 106
  LH Week 48 | 0.367 (8.5631)
  LH Week 72: number analyzed (Participants) | 23
  LH Week 72 | 0.222 (6.8910)

20. Secondary Outcome: Gonadal (FSH and LH) Hormone Values for Male Participants From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: SAF (Male participants who received any study drug); Here, "Number Analyzed" = Number of male participants evaluable at that timepoint
Measure: Mean (Standard Deviation); unit: International units per litre (IU/L)
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 858
International units per litre (IU/L)
  FSH Baseline | 8.006 (7.4451)
  FSH Week 8: number analyzed (Participants) | 117
  FSH Week 8 | 7.959 (7.5500)
  FSH Week 12: number analyzed (Participants) | 215
  FSH Week 12 | 7.766 (6.8204)
  FSH Week 24: number analyzed (Participants) | 489
  FSH Week 24 | 8.268 (8.1355)
  FSH Week 48: number analyzed (Participants) | 203
  FSH Week 48 | 9.597 (11.2138)
  FSH Week 72: number analyzed (Participants) | 32
  FSH Week 72 | 10.005 (13.2973)
  LH Baseline | 6.500 (4.2832)
  LH Week 8: number analyzed (Participants) | 117
  LH Week 8 | 7.094 (4.7226)
  LH Week 12: number analyzed (Participants) | 215
  LH Week 12 | 6.688 (4.4079)
  LH Week 24: number analyzed (Participants) | 489
  LH Week 24 | 6.931 (4.8597)
  LH Week 48: number analyzed (Participants) | 203
  LH Week 48 | 7.677 (6.5478)
  LH Week 72: number analyzed (Participants) | 32
  LH Week 72 | 8.173 (8.9083)

21. Secondary Outcome: Change From Baseline in Gonadal Hormones (FSH and LH) for Male Participants Over Time
Time Frame: Up to week 72
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 858
IU/L
  FSH Week 8: number analyzed (Participants) | 117
  FSH Week 8 | 0.285 (3.7264)
  FSH Week 12: number analyzed (Participants) | 215
  FSH Week 12 | -0.598 (4.1076)
  FSH Week 24: number analyzed (Participants) | 489
  FSH Week 24 | 0.331 (6.0522)
  FSH Week 48: number analyzed (Participants) | 203
  FSH Week 48 | 0.960 (10.3803)
  FSH Week 72: number analyzed (Participants) | 32
  FSH Week 72 | 2.458 (13.4730)
  LH Week 8: number analyzed (Participants) | 117
  LH Week 8 | 0.535 (2.4847)
  LH Week 12: number analyzed (Participants) | 215
  LH Week 12 | -0.136 (3.2638)
  LH Week 24: number analyzed (Participants) | 489
  LH Week 24 | 0.582 (4.4964)
  LH Week 48: number analyzed (Participants) | 203
  LH Week 48 | 1.015 (6.6344)
  LH Week 72: number analyzed (Participants) | 32
  LH Week 72 | 1.964 (9.3028)

22. Secondary Outcome: Gonadotropin (Estradiol) Values for Female Participants From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: picomoles per litre (pmol/L)
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 527
picomoles per litre (pmol/L)
  Baseline | 55.589 (80.8238)
  Week 8: number analyzed (Participants) | 84
  Week 8 | 58.676 (69.0119)
  Week 12: number analyzed (Participants) | 135
  Week 12 | 59.673 (74.7587)
  Week 24: number analyzed (Participants) | 280
  Week 24 | 64.304 (103.8955)
  Week 48: number analyzed (Participants) | 106
  Week 48 | 64.503 (102.1595)
  Week 72: number analyzed (Participants) | 23
  Week 72 | 57.926 (67.1795)

23. Secondary Outcome: Change From Baseline in Gonadotropins (Estradiol) for Female Participants Over Time
Time Frame: Up to week 72
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 527
pmol/L
  Week 8: number analyzed (Participants) | 84
  Week 8 | 4.272 (77.1561)
  Week 12: number analyzed (Participants) | 135
  Week 12 | 9.262 (73.1050)
  Week 24: number analyzed (Participants) | 280
  Week 24 | 7.869 (78.4151)
  Week 48: number analyzed (Participants) | 106
  Week 48 | 11.763 (97.5350)
  Week 72: number analyzed (Participants) | 23
  Week 72 | 9.569 (38.0952)

24. Secondary Outcome: Gonadotropin (Testosterone) Values for Male Participants From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: nanomoles per litre (nmol/L)
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 858
nanomoles per litre (nmol/L)
  Baseline | 13.4370 (6.36321)
  Week 8: number analyzed (Participants) | 117
  Week 8 | 14.5802 (5.99821)
  Week 12: number analyzed (Participants) | 215
  Week 12 | 14.2443 (6.77070)
  Week 24: number analyzed (Participants) | 489
  Week 24 | 13.5818 (6.11269)
  Week 48: number analyzed (Participants) | 203
  Week 48 | 13.4798 (7.04977)
  Week 72: number analyzed (Participants) | 32
  Week 72 | 12.7538 (6.37408)

25. Secondary Outcome: Change From Baseline in Gonadotropins (Testosterone) for Male Participants Over Time
Time Frame: Up to week 72
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 858
nmol/L
  Week 8: number analyzed (Participants) | 117
  Week 8 | 0.6030 (4.46401)
  Week 12: number analyzed (Participants) | 215
  Week 12 | 0.7965 (4.74765)
  Week 24: number analyzed (Participants) | 489
  Week 24 | 0.1946 (5.89220)
  Week 48: number analyzed (Participants) | 203
  Week 48 | 0.0498 (6.34201)
  Week 72: number analyzed (Participants) | 32
  Week 72 | 1.2569 (5.29335)

26. Secondary Outcome: Alanine Aminotransferase Values From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L (Units per Liter)
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
U/L (Units per Liter)
  Baseline | 0.516 (0.3218)
  Week 8: number analyzed (Participants) | 201
  Week 8 | 0.468 (0.2745)
  Week 12: number analyzed (Participants) | 350
  Week 12 | 0.505 (0.4940)
  Week 24: number analyzed (Participants) | 769
  Week 24 | 0.493 (0.2851)
  Week 48: number analyzed (Participants) | 310
  Week 48 | 0.533 (0.3267)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 0.468 (0.2340)

27. Secondary Outcome: Change From Baseline in Alanine Aminotransferase Over Time
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
U/L
  Week 8: number analyzed (Participants) | 201
  Week 8 | -0.025 (0.3006)
  Week 12: number analyzed (Participants) | 350
  Week 12 | 0.009 (0.5189)
  Week 24: number analyzed (Participants) | 769
  Week 24 | -0.036 (0.3294)
  Week 48: number analyzed (Participants) | 310
  Week 48 | -0.027 (0.3052)
  Week 72: number analyzed (Participants) | 54
  Week 72 | -0.062 (0.1872)

28. Secondary Outcome: Aspartate Aminotransferase Values From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
U/L
  Baseline | 0.553 (0.2516)
  Week 8: number analyzed (Participants) | 201
  Week 8 | 0.520 (0.2536)
  Week 12: number analyzed (Participants) | 350
  Week 12 | 0.527 (0.2698)
  Week 24: number analyzed (Participants) | 769
  Week 24 | 0.544 (0.3071)
  Week 48: number analyzed (Participants) | 310
  Week 48 | 0.565 (0.2773)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 0.556 (0.2256)

29. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase Over Time
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
U/L
  Week 8: number analyzed (Participants) | 201
  Week 8 | -0.022 (0.2856)
  Week 12: number analyzed (Participants) | 350
  Week 12 | -0.017 (0.3004)
  Week 24: number analyzed (Participants) | 769
  Week 24 | -0.013 (0.2901)
  Week 48: number analyzed (Participants) | 310
  Week 48 | -0.019 (0.2390)
  Week 72: number analyzed (Participants) | 54
  Week 72 | -0.037 (0.1730)

30. Secondary Outcome: Alkaline Phosphatase Values From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
U/L
  Baseline | 0.601 (0.1865)
  Week 8: number analyzed (Participants) | 201
  Week 8 | 0.635 (0.2151)
  Week 12: number analyzed (Participants) | 350
  Week 12 | 0.605 (0.1865)
  Week 24: number analyzed (Participants) | 769
  Week 24 | 0.602 (0.2012)
  Week 48: number analyzed (Participants) | 310
  Week 48 | 0.602 (0.2657)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 0.553 (0.1678)

31. Secondary Outcome: Change From Baseline in Alkaline Phosphatase Over Time
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
U/L
  Week 8: number analyzed (Participants) | 201
  Week 8 | 0.009 (0.1371)
  Week 12: number analyzed (Participants) | 350
  Week 12 | 0.013 (0.1203)
  Week 24: number analyzed (Participants) | 769
  Week 24 | 0.006 (0.1152)
  Week 48: number analyzed (Participants) | 310
  Week 48 | 0.024 (0.2333)
  Week 72: number analyzed (Participants) | 54
  Week 72 | -0.011 (0.1029)

32. Secondary Outcome: Total Bilirubin Values From Baseline Over Time
Description: as for outcome 2
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micromoles per litre (umol/L)
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
micromoles per litre (umol/L)
  Baseline | 10.76 (4.736)
  Week 8: number analyzed (Participants) | 201
  Week 8 | 10.01 (4.123)
  Week 12: number analyzed (Participants) | 350
  Week 12 | 10.26 (4.758)
  Week 24: number analyzed (Participants) | 769
  Week 24 | 10.41 (4.922)
  Week 48: number analyzed (Participants) | 310
  Week 48 | 10.06 (4.503)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 8.82 (3.770)

33. Secondary Outcome: Change From Baseline in Total Bilirubin Over Time
Time Frame: Up to week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
Number analyzed (Participants) | 1385
umol/L
  Week 8: number analyzed (Participants) | 201
  Week 8 | -0.37 (3.120)
  Week 12: number analyzed (Participants) | 350
  Week 12 | -0.44 (3.854)
  Week 24: number analyzed (Participants) | 769
  Week 24 | -0.48 (3.962)
  Week 48: number analyzed (Participants) | 310
  Week 48 | -0.05 (3.991)
  Week 72: number analyzed (Participants) | 54
  Week 72 | 0.71 (2.152)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of signed informed consent until the end of study, up to 80 weeks.
Description: Treatment-emergent adverse events (TEAEs) are reported. TEAEs are AEs that developed or worsened or became serious during the TEAE period (time from first dose of study drug to the last study visit).
Arm/Group | Alirocumab 75 Q2W/Up150 Q2W
All-Cause Mortality (participants affected / at risk) | 5/1385
Serious Adverse Events (participants affected / at risk) | 89/1385
Other Adverse Events (participants affected / at risk) | 0/1385
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alirocumab 75 Q2W/Up150 Q2W (N=1385)
Angina unstable (Cardiac disorders) | 10 (10)
Angina pectoris (Cardiac disorders) | 8 (8)
Atrial fibrillation (Cardiac disorders) | 6 (6)
Acute myocardial infarction (Cardiac disorders) | 5 (5)
Acute left ventricular failure (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Abscess limb (Infections and infestations) | 1 (1)
Appendiceal abscess (Infections and infestations) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 2 (2)
Carotid artery disease (Nervous system disorders) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1)
Chest pain (General disorders) | 3 (3)
Death (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Electric shock (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Synovial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (2)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Cataract (Eye disorders) | 1 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT03694197/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT03694197/SAP_001.pdf